CLINICAL TRIAL: NCT00121368
Title: Survey on Tobacco Use in the GN Sites
Brief Title: GN Tobacco Use Survey
Status: Completed | Type: Observational
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); RTI International (Other)
Responsible Party: Sponsor
Other Study IDs: CP01 Tobacco Use
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Smoking
Keywords: Global Network; Maternal and child health; International; Women's health; Tobacco; Smoking; Africa; Latin America; South America; Guatemala; Zambia; India; Argentina; Democratic Republic of the Congo
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Smoking can contribute to many health problems for mothers and their babies. In developing countries, there is little information about the number of pregnant women that smoke and the reasons why some pregnant women choose to smoke. The purpose of this multi-site tobacco use survey is to obtain information on knowledge, attitudes and behaviors among pregnant women in diverse populations regarding tobacco products.

DETAILED DESCRIPTION:
Smoking is regarded as one of the few potentially preventable factors associated with low birth weight, very preterm birth and perinatal death. In an effort to determine the prevalence of tobacco use (smoking and smokeless tobacco) and to collect relevant data in support of a potential smoking prevention or cessation intervention, a multi-site tobacco use survey is being conducted in several countries. The survey will be used to obtain information on knowledge, attitudes and behaviors among pregnant women in diverse populations regarding tobacco products.

The primary outcome is tobacco use status during pregnancy. Secondary outcomes include: knowledge and attitudes regarding tobacco products, health hazards of tobacco use and environmental tobacco smoke (ETS) exposure.

Sample size of 750 per country was calculated under the assumptions that the prevalence of tobacco use could be as low as 0.05 with a coefficient of variation of approximately 15% and a prevalence of 0.10 with a CV of approximately 11%.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of legal consent and child-bearing age (18-45)
* Attendance at a participating clinic

Exclusion Criteria:

* Pregnant women with disabilities such as deafness, serious mental illness, or mental retardation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women 18-45
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Actual)
Dates: Start 2004-02; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Tobacco use | Cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Michele Bloch, MD, PhD, Principal Investigator — National Cancer Institute (NCI)
Locations (9):
- Buenos Aires, Argentina
- Recife, Brazil
- Quito, Ecuador
- Guatemala City, Guatemala
- India (2):
  - Bhubaneswar, Odisha
  - Belagavi
- Karachi, Pakistan
- Kinshasa, Republic of the Congo
- Lusaka, Zambia

REFERENCES:
- See also: Global Network for Women's and Children's Health — http://gn.rti.org/